CLINICAL TRIAL: NCT06513182
Title: Do Wound Protectors Reduce Contamination in Total Shoulder Arthroplasty? A Randomized Controlled Trial
Brief Title: Do Wound Protectors Reduce Contamination in Total Shoulder Arthroplasty?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Joyce, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 179068
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Cutibacterium Acnes
Keywords: Total shoulder arthroplasty; Wound protector; Cutibacterium acnes; Contamination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control - no wound protector (Other): The (control - no wound protector) will not use the protector device during the course of the surgery. During surgery 4 tissue swab cultures will be obtained and sent to a laboratory for analysis.
  Interventions: Other: No Alexis orthopaedic protector
- Wound protector (Experimental): Wound protector group will have an insertion of a wound protector after making an initial superficial approach to the shoulder. During surgery 4 tissue swab cultures will be obtained and sent to a laboratory for analysis. The wound protector will then remain in place until the end of the case during wound closure.
  Interventions: Device: Alexis orthopaedic protector

INTERVENTIONS:
Other: No Alexis orthopaedic protector — No Alexis orthopaedic protector will be used during the course of the surgery.
  Arms: Control - no wound protector
Device: Alexis orthopaedic protector — Alexis orthopaedic protector will be inserted after making an initial superficial approach to the shoulder.
  Other Names: Wound protector; Rigid Retraction Ring; Flexible Retraction Ring
  Arms: Wound protector

SUMMARY:
Prosthetic joint infection is a devastating complication of shoulder arthroplasty. A relatively novel method of preventing PJI has been with the use of a wound protection device. There is minimal investigative research on the use of a wound protector in shoulder arthroplasty, specifically with an ability to decrease wound contamination. The investigators primary purpose of the proposed study is to determine if the use of a wound protector deceases the deep wound colonization of bacteria in primary shoulder arthroplasty. A secondary purpose is to evaluate if the wound protector decreases soft tissue trauma during total shoulder arthroplasty.

DETAILED DESCRIPTION:
Prosthetic joint infection (PJI) is a relatively uncommon but devastating complication of shoulder arthroplasty. Published rates of PJI after shoulder arthroplasty range one to ten percent. Since the advent of surgery, infection has been a constant battle. As a profession, we have made strides in preventing infection. Infection prevention started with the popularization of hand washing and preparation and draping of the sterile field in the nineteenth and twentieth centuries, with more recent advancements including pre-operative and intra-operative antimicrobial washes, antibiotic powders, and ultraviolent light exposure. Despite these advancement, PJI continues to be a problem in orthopaedic arthroplasty surgery, and we need to continue to improve our infection prevention techniques.

Risk factors for PJI in shoulder arthroplasty include revision surgery, obesity, male gender, younger age, and non-osteoarthritis indication for surgery. Unfortunately, the majority of these risk factors are non-modifiable and are difficult to mitigate short of avoiding surgery on these patients. Due to this, surgeons need to continue to find ways of preventing PJI both pre-operatively and intra-operatively. The most frequent bacteria responsible for shoulder PJI are cutibacterium acnes and s. epidermidis, causing an estimated 67 and 27 percent of shoulder PJIs respectively. C. acnes is difficult to prevent due to its prevalence in the sebaceous glands in the shoulder, neck, and upper back area. Published methods of preventing c. acnes infection include pre-operative antibiotics, skin preparation with hydrogen peroxide wash, betadine wash after skin incision, and many others. Most of these methods focus on destroying the bacterium that are present in the wound. The inherent problem is that c. acnes is symbiotic and lives in human skin, therefore attempting to destroy it is an uphill battle as it will continue to recolonize the wound through the operation.

A relatively novel method of preventing PJI has been with the use of a wound protection device. While there is some outcome data with the use of this device in hip arthroplasty, there is minimal data in regards to shoulder arthroplasty. The only peer-reviewed study of use of a flexible wound protector in shoulder arthroplasty demonstrated a decrease in c. acnes colonization in shoulder wounds after placement of a wound protector. The purpose of the proposed study is to determine if the use of a wound protector deceases the deep wound colonization of c. acnes in primary shoulder arthroplasty.

PRELIMINARY STUDIES:

A study at the investigators institution looked at the use of a hydrogen peroxide skin preparation prior to shoulder arthroplasty surgery, and found that the standardized peroxide preparation decreased surgical wound colonization with c. acnes to 10 percent versus 35 percent in the control group. While the proposed study is different, the investigators intend to use a similar study protocol as this is a proven protocol that worked effectively within this institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary anatomic or reverse shoulder arthroplasty by one of three surgeons will be eligible.

Exclusion Criteria:

* revision arthroplasty,
* history of ipsilateral shoulder infection,
* patients unable or unwilling to consent,
* prisoners,
* pregnant individuals,
* mentally disabled patients,
* employees of the University of Utah,
* allergy to polyurethane polyester.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Positive C acnes culture | 2-weeks
  The primary outcome of the study will be percent of positive C acnes culture results.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Joyce, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No